CLINICAL TRIAL: NCT03557996
Title: Discoloration of Carious Primary Teeth After Application of Silver Diamine Fluoride Versus Sodium Fluoride Varnish: A Randomized Clinical Trial
Brief Title: Discoloration of Carious Primary Teeth After Application of Silver Diamine Fluoride Versus Sodium Fluoride Varnish
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yousra Mohamed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-06-2
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Dental Caries in Children
MeSH Terms: interventions — silver diamine fluoride; Bifluorid 12

STUDY DESIGN:
Intervention Model Description: patient will receive either silver diamine fluoride or sodium fluoride varnish
Who Masked: Participant, Outcomes Assessor
Masking Description: double (participant-outcome assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 (Experimental): 38% silver diamine fluoride liquid will be applied twice annually and patients will be followed up as 0,1,3,6,9 and 12 SDF is brush on liquid
  Interventions: Drug: Silver Diamine Fluoride
- Group 2 (Active Comparator): 5% Sodium fluoride varnish will be applied four times annually and patient will be followed up at 0,1,3,6,9 and 12
  Interventions: Drug: Sodium Fluoride Varnish

INTERVENTIONS:
Drug: Silver Diamine Fluoride — SDF will be applied with a brush
  Other Names: SDF
  Arms: Group 1
Drug: Sodium Fluoride Varnish — NaF will be applied with a brush
  Other Names: NaF varnish
  Arms: Group 2

SUMMARY:
To assess discoloration of carious primary teeth after application of silver diamine fluoride versus sodium fluoride varnish.

DETAILED DESCRIPTION:
The American Academy of Pediatric Dentistry's (AAPD) guidelines (2017) stated that Silver diamine fluoride (SDF) is a brush-on liquid that arrest 87.7% of dental caries lesions. The success rate is similar for restorations placed under GA. One of the most exciting aspects of SDF is the 67±4% decrease in new lesions on untreated surfaces, achieved simply by treating active lesions .This is not the same as incidence of any new lesions (elaborated above for treatment under GA), however the relation warrants further investigation.

Benefit to the patient

* No pain and infection.
* Enhance child cooperation.
* Enhance better patient compliance.
* Decrease cost of dental treatment and may eliminate the need for General Anesthesia.

Benefit to the dentist

* Develop an effective fast easy method to arrest the caries by using SDF.
* Ease of dental treatment.
* Better cooperation with the child.
* The procedure is simple.
* Inexpensive and non-invasive.
* It does not require expensive equipment or support infrastructure, such as pipe water or electricity.

Benefit to the population

* Reduce the harmful impact of oral health problems in preschool children from low income families.
* SDF can be considered a user-friendly material for use in dental clinics as well as remote areas, schools or deprived communities.

Children aged 2-5 years can benefit from the use of SDF, an easy anticaries treatment. Furthermore, children in this age group may benefit from delayed dental treatment and overall caries arrest, thus reducing potential pain and infection, expensive future emergency room visits, the need for general anesthesia or traumatic dental experiences on uncooperative children.

ELIGIBILITY:
Inclusion Criteria:

1. Children with carious primary teeth before eruption of permanent teeth
2. High caries risk patients with anterior or posterior carious lesions
3. Uncooperative children without access to or with difficulty accessing dental care.

Exclusion Criteria:

1. Children with spontaneous or elicited pain from caries
2. Tooth mobility
3. Signs of pulpal infection
4. Severe medical conditions that would not allow management in the clinic

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Discoloration | 12 months
  Discoloration will be assessed by questioning the patient and/or the guardian.binary (yes or no)

SECONDARY OUTCOMES:
Investigator reported discoloration | 12 months
  Investigator will report the discoloration occurred to treated teeth (yellow, brown, black) Visual examination
Timing of discoloration | 12 months
  Visual examination at follow up
Caries arrest (dentine texture) | 12 months
  Caries arrest will be assessed through tactile examination (Soft or hard) Tactile examination
Postoperative Pain: Questioning the patient | 12 months
  Questioning the patient and/or the parentBinary (yes or No)
Parental satisfaction: Questioning the parent | 12 months
  Questioning the parent

CONTACTS AND LOCATIONS:
Overall Officials: Nevine G Waly, Professor, Study Director — Pediatric Dentistry,Faculty of Dentistry, Cairo University; Eman S Elmasry, Professor, Study Chair — Pediatric Dentistry, Faculty of Dentistry, Cairo University; Fatma KI Abdelgawad, Lecturer, Study Director — Pediatric Dentistry, Faculty of Dentistry, Cairo University; Yousra M Abdel Rehim, MSc, Principal Investigator — Pediatric Dentistry, Faculty of Dentistry, Cairo University
Locations (1):
- Pediatric Dentistry, Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
outcome results for both groups will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: to be determined later
Access Criteria: to be determined later